CLINICAL TRIAL: NCT06107166
Title: Testosterone and Vascular Function in Reproductive-Aged Females With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Sandra Dumanski, Assistant Professor, University of Calgary
Other Study IDs: REB18-0642
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death among women and women with chronic kidney disease are at an even greater risk of CVD. The aim of this observational study is to examine the relationship between total testosterone levels and measures of vascular function (pulse wave velocity, aortic augmentation index, flow mediated dilation and velocity time integral) in reproductive-aged women living with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* a diagnosis of chronic kidney disease or end stage kidney disease
* age 18-51

Exclusion Criteria:

Pregnancy, breastfeeding, current use of menopausal hormone therapy or gender affirming hormone therapy, or factors that would affect ovarian function, such as polycystic ovarian syndrome, premature ovarian insufficiency, ovarian malignancy, gonadotoxic chemotherapy, surgical oophorectomy, or previous radiation to the pelvis.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will include stable females of reproductive age (18-51 years of age) with chronic kidney disease. Subjects will require permission of their primary nephrologist or primary care provider to participate
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity | Measured at baseline
Aortic augmentation index | Measured at baseline
Flow mediated dilation | Measured at baseline
Velocity time integral | Measured at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No